CLINICAL TRIAL: NCT06636331
Title: Comparison of The Continous Suprainguinal Fascia Iliaca Compartment Block and Continous Epidual on The Quality of Postoperative Analgesia, Interleukin-6, Hemodynamic Stability and QoR-40 for Cephalomedullary Nailing Surgeries
Brief Title: Comparison of The Continous Suprainguinal Fascia Iliaca Compartment Block and Continous Epidural
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Riko, MD, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Udayana University
Record Dates: First submitted 2024-10-06; First posted 2024-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative
Keywords: Pain Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment S-FICB Arm (Experimental): S-FICB with PCRA using Ropivacaine 0.2% continuous 2ml/hr, demand dose 5ml as needed.
  Interventions: Other: Continuous Suprainguinal Fascia Iliaca Compartment Block
- Treatment Epidural Arm (Experimental): Epidural with PCEA using Ropivacaine 0.2% continuous 2ml/hr, demand dose 5ml as needed.
  Interventions: Other: Continuous Epidural

INTERVENTIONS:
Other: Continuous Suprainguinal Fascia Iliaca Compartment Block — Using PCRA and Local Anesthetic Ropivacaine 0.2% continuous 2ml/hr and demand dose 5ml as needed.
  Arms: Treatment S-FICB Arm
Other: Continuous Epidural — Using PCEA and Local Anesthetic Ropivacaine 0.2% continuous 2ml/hr and demand dose 5ml as needed.
  Arms: Treatment Epidural Arm

SUMMARY:
This study evaluates the effectiveness of postoperative analgesia quality, Interleukin-6, Hemodynamic stability and QoR-40 of continuous Suprainguinal Fascia Iliaca Compartment Block (S-FICB) compared with continuous epidural in patients undergoing cephalomedullary nailing surgery.

Half of participants will receive continuous S-FICB with patient control regional analgesia using ropivacaine 0.2% continue 2ml/hr and demand dose 5ml as needed, while the other half will receive continuous epidural with patient control epidural analgesia using same regimen.

DETAILED DESCRIPTION:
The Continuous Suprainguinal Fascia Iliaca Compartment Block (S-FICB) and continuous epidural are regional anaesthesia that can be used to relieve postoperative pain of femur surgery. But there are few studies have been done to compare both techniques.

The S-FICB is an alternate peripheral nerve block technique using local anaesthetic administered into the fascia iliaca compartment at the inguinal region which targets the femoral, obturator and lateral femoral cutaneous nerves.

The epidural is well known and proven to have an adequate analgesia effect using local anaesthetic in the epidural region targeted for femur surgery.

Based on previous studies, the effectiveness of the S-FICB single shot was no longer than 18 hours. Then we choose to continue S-FICB to find out how adequate it is. The S-FICB with ropivacaine has a proven anti-inflammatory effect for the first 24 hours postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients is planned for cephalomedullary nailing surgery
2. Patients with BMI 18 - 30 kg/m2
3. Patients with ASA physical status I - III

Exclusion Criteria:

1. Patients with contraindications to regional anesthesia
2. Patients with mental disorders or psychiatric disorders
3. Patients have a history of allergy to the local anesthetic drug
4. Patients or family refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
The Quality of Postoperative Analgesia | 24 hours
  Assess the local anesthetic dosage in milligrams from patient controlled analgesia Machine for attempt dose, delivered dose and 24 hours total doses.

SECONDARY OUTCOMES:
Delta Interleukin-6 | 3 days
  Laboratory report for interleukin-6 preoperative and 24 hours posoperative then calculate the delta Interleukin-6
Hemodynamic Stability | 24 hours
  Monitoring blood pressure category as stable or not stable. Stable if systolic blood pressure is above 100 mmHg. Not Stable if systolic blood pressure is under 100 mmHg.
Questionnaire of Recovery 40 (QoR-40) | 24 hours
  Assess the subject recovery condition using questionnaires QoR-40. The score range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Tjokorda Gde Agung Senapathi, Principal Investigator — Udayana University; I Gusti Ngurah Mahaalit Aribawa, Principal Investigator — Udayana University; I Gusti Agung Gede Utara Hartawan, Principal Investigator — Udayana University; I Gede Budiartha, Principal Investigator — Udayana University; I Made Gede Widnyana, Principal Investigator — Udayana University; Made Agus Kresna Sucandra, Study Chair — Udayana University; Ida Bagus Krisna Jaya Sutawan, Study Chair — Udayana University; I Putu Pramana Suarjaya, Study Chair — Udayana University
Locations (2):
- Indonesia (2):
  - Prof IGNG Ngoerah Hospitals, Denpasar, Bali
  - Udayana University, Denpasar, Bali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Sherbeny, S., Maguid, H., El Dourgham, L., Ibrahim, O., Patient Controlled Analgesia: Fascia Iliaca Compartment Block Versus Epidural Analgesia for Postoperative Pain Relief Following Total Knee Replacement Under Spinal Anesthesia: A Comparative Study. Zagazig University Medical Journal, 2022; (318-325): -.doi: 10.21608/zumj.2020.28085.1821
- [Background] Azizoglu M, Rumeli S. Comparison of the suprainguinal fascia iliaca compartment block with continuous epidural analgesia in patients undergoing hip surgeries: a retrospective study. Braz J Anesthesiol. 2022 May-Jun;72(3):342-349. doi: 10.1016/j.bjane.2021.07.006. Epub 2021 Jul 26. PMID 34324929
- [Background] Zhu K, Zheng F, Wang C, Ding L. Effect of Ultrasound-Guided Fascia Iliac Compartment Block on Serum NLRP3 and Inflammatory Factors in Patients with Femoral Intertrochanteric Fracture. Comput Math Methods Med. 2022 May 17;2022:1944659. doi: 10.1155/2022/1944659. eCollection 2022. PMID 35620203
- See also: The World Federation of Societies of Anaesthesiologists have updated information about Fascia Iliaca Compartment Block — https://resources.wfsahq.org/atotw/fascia-iliaca-compartment-block-an-update/